CLINICAL TRIAL: NCT05124873
Title: Moisture Management Liner At-Home Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturing delays and issues of the experimental liner due to the Covid-19 pandemic. Manufacturers unable to provide the remaining liners to the investigators in the required timeframe.
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Vivonics, Inc. (Industry)
Responsible Party: Principal Investigator, Todd Farrell, Director of Research, Liberating Technologies, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E00572.2a; 2020/09/1 (Other: Solutions IRB); E00572.2b (Other: HRPO)
Record Dates: First submitted 2021-06-28; First posted 2021-11-18 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Amputation Stump; Amputation; Amputees; Lower Limb Deformity; Prosthesis User; Prosthesis
Keywords: Cooling; amputee; lower limb difference; Prosthetic; socket; Prosthesis; Prosthetist; Liner; sweat; walking; sock; leg; perspiration; moisture; heat; thermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Prosthetic Liner (Experimental): Moisture Management Liner: A prototype liner designed to reduce heat that builds up on the limb. The participant wears this liner at home for about 4 weeks and provides feedback on the prototype.
  Interventions: Device: Moisture Management Liner

INTERVENTIONS:
Device: Moisture Management Liner — A prototype liner designed to reduce heat that builds up on the limb.

SUMMARY:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by unbreathable and non-thermally conductive materials that can create a warm and ultimately moist environment.

The investigators have developed a silicone liner approach to passively conduct heat from the skin using thermally conductive elastomers. A technology that can provide thermal control while retaining adequate suspension, weight, and other prosthetic characteristics would benefit many prosthesis wearers.

DETAILED DESCRIPTION:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by unbreathable and non-thermally conductive materials that can create a warm and ultimately moist environment. These layers consist of a prosthetic liner that rolls onto the limb and traps heat and occasional extra prosthetic socks. Studies found increases in socket temperature after the prosthesis was donned. Temperatures were found to remain elevated long after activity cessation and even a rest period of double the duration of the preceding activity period is insufficient to return the limb to its initial temperature. A small amount of activity can cause the socket temperature to elevate and remain at an uncomfortable level for an extended period of time, which can lead to decreased wear times. In summary, an uncomfortable socket/residual limb interface decreases prosthesis use among amputees who want to remain active in their lives.

The investigators have developed a silicone liner approach to passively conduct heat from the skin using thermally conductive elastomers. A technology that can provide thermal control while retaining adequate suspension, weight, and other prosthetic characteristics would benefit many prosthesis wearers.

This study will focus on investigating the efficacy of this novel moisture and thermal management (experimental) liner.

The rationale for this study is to determine how well the new technology can regulate the residual limb temperature and reduce the moisture generation in a home environment where the device would ultimately be utilized.

The objective of this study is to measure the effects of residual limb moisture and thermal management on quality of life (QoL) and functional outcomes. Reducing temperature increases of the residual limb inside the prosthetic socket would result in less sweating and greater comfort while wearing the prosthesis, and ultimately greater function and better quality of life as measured by standard functional and QoL outcome measures. The primary outcome measure is the modified Dermatology Quality Life Index (mDLQI). All other measures collected during this study are exploratory.

A prospective design will be implemented for this study. Research participants will be consented by LTI over the phone. Residual limb measurements will be received from the participant to confirm liner sizing. One 'experimental' prototype liner will be created for each participant. Subjects with a similar liner size and profile to the available experimental liners will be targeted. Temperature and step-count sensors will be placed on the participant's prosthesis to log daily measurements. Testing will consist of 2 site visits, with the entire study lasting approximately 5 weeks.

Lower limb prosthesis users will be recruited for the study and consented with an approved protocol. Research participants will represent a convenience sample and will reflect the local population of people with lower limb differences who use prosthetic sockets and could benefit from temperature control within the socket.

A maximum of 16 subjects will be recruited for this study. This sample size accounts for subject drop out and other losses (such as incomplete log data, etc.) to yield usable data from the target 12 subjects required by the power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputee
* Be willing and able to complete the tasks outlined
* Are at least 6 months on a lower-limb prosthesis
* Fits within an experimental liner (cushion style liner and size 23.5-28 cm)
* Can understand English in order to be properly consented and provide their feedback to the study personnel

Exclusion Criteria:

* The risks to pregnant women and fetuses are unknown and therefore pregnant women should not participate in the study
* Other unforeseen disqualifying criteria (such as specific cognitive issues, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Liberating Technologies, Inc., Holliston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Prosthetic Liner
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Prosthetic Liner
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1
Modified Dermatology Life Quality Index (mDLQI) [Number; unit: units on a scale] — The modified Dermatology Life Quality Index (mDLQI) is a modified version of the Dermatology Life Quality Index (DLQI). The DLQI is a simple questionnaire designed to measure the health-related quality of life of adult patients suffering from various skin diseases. A modified version of the questionnaire (mDLQI) was developed to be more directly applicable to persons with amputation (i.e., revised wording to apply to the skin on their residual limb). The modified survey is scored from 0 to 27, with lower numbers indicating a better outcome.
  units on a scale | 5

OUTCOME MEASURES:

1. Primary Outcome: Modified Dermatology Life Quality Index (mDLQI)
Description: The modified Dermatology Life Quality Index (mDLQI) is a modified version of the Dermatology Life Quality Index (DLQI). The DLQI is a simple questionnaire designed to measure the health-related quality of life of adult patients suffering from various skin diseases. A modified version of the questionnaire (mDLQI) was developed to be more directly applicable to persons with amputation (i.e., revised wording to apply to the skin on their residual limb). The modified survey is scored from 0 to 27, with lower numbers indicating a better outcome.
Time Frame: 4 weeks
Measure: Number; unit: units on a scale
Arm/Group | Experimental Prosthetic Liner
Number analyzed (Participants) | 1
units on a scale | 7

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/collected during the entire study (about 5 weeks). Participants were told to reach out to study staff immediately if adverse events did occur.
Arm/Group | Experimental Prosthetic Liner
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05124873/Prot_SAP_000.pdf